CLINICAL TRIAL: NCT02320279
Title: The Fetal EKG Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mindchild Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: South Shore Fetal EKG study
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Labor
Keywords: Fetal Heart Rate; Fetal EKG; FHR tracing; fetal R-waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women in labor: Pregnant women, women in labor, and women who are admitted to labor and delivery for scheduled c-sections will form the eligible population for recruitment into our study.
  Interventions: Device: Fetal Heart Rate Monitor

INTERVENTIONS:
Device: Fetal Heart Rate Monitor — Use of a system that monitors fetal heart rate through use of fetal EKG read using abdominal electrodes
  Other Names: Mindchild Meridian Fetal Heart Rate System

SUMMARY:
The objective is to contribute data to ongoing research activities focused on identification of EKG waveform changes in the context of clinical conditions and maternal medication use. Additionally, to develop the capacity to measure contractions more accurately and more reliably using skin-surface electrodes.

DETAILED DESCRIPTION:
Specific Aim 1: To develop a technique for the quantitative analysis of fetal heart-rate (FHR) data recorded during labor using advanced mathematical techniques, including pattern-recognition analysis.

* Specific Aim 2: To develop the capacity to measure fetal cardiac data using EKG sensors applied to the maternal abdomen during labor.
* Specific Aim 3: To validate prenatal non-invasive measurement of the fetal QTc interval.
* Specific Aim 4: To develop and validate the capacity to measure uterine contractions using the uterine EMG signal recorded from maternal skin-surface electrodes.
* Specific Aim 5: Collect clinical data related to medication usage and hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant or in labor who are having their fetus' heart rate monitored continuously and able to consent
* 18 years old or older.
* Gestational age of 24-42 weeks.
* Any method of fetal heart rate monitoring.
* Pregnant women in labor as well as women who are not in labor.
* Pregnant women who are admitted to labor and delivery for scheduled c-sections.

Exclusion Criteria:

* Women unable to consent
* Women under sedation or systemic anesthesia, and women who have diminished cognitive capacity
* Women in extremis (in severe pain, etc.)
* Women who are using the Mindchild device for clinical monitoring.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, women in labor, and women who are admitted to labor and delivery for scheduled c-sections will form the eligible population for recruitment into our study. These women will be identified by a study staff-member who will ask on-call physicians, midwives, and nurses working on Labor and Delivery
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2013-10; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative FHR | During Labor
  Quantitative analysis of fetal heart-rate data recorded during labor using advanced mathetmatical techniques, including pattern-recognition analysis using EKG electrodes applied to the maternal abdomen.

SECONDARY OUTCOMES:
Uterine contractions | During labor
  Uterine contractions will be identified by analyzing data from surface electrodes to identify patterns consistent with uterine muscle coordinated shortening. These data will be compared to data from either the external tocometer or the internal IUPC. Cross correlation analysis will be used to compare the two signals and validate the analysis of uterine EMG signal.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wolfberg, MD, Principal Investigator — South Shore Hospital
Locations (1):
- South Shore Hospital, South Weymouth, Massachusetts, United States